CLINICAL TRIAL: NCT00107835
Title: An Open-Label Safety Study to Evaluate the Use of S-Caine™ Peel (Lidocaine 7% and Tetracaine 7% Cream) in Adult Patients Undergoing a Minor or Major Dermal Procedure
Brief Title: Safety Study of S-Caine Peel (Skin Numbing Cream) Before a Painful Dermatologic Procedure in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ZARS Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCP-45-05
Record Dates: First submitted 2005-04-08; First posted 2005-04-11 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Pain
Keywords: Pain
MeSH Terms: conditions — Pain | interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- S-Caine Peel (Experimental)
  Interventions: Drug: S-Caine™ Peel (lidocaine and tetracaine cream 7%/7%)

INTERVENTIONS:
Drug: S-Caine™ Peel (lidocaine and tetracaine cream 7%/7%) — S-Caine Peel comprising a 1:1 eutectic mixture of 7% lidocaine, and 7% tetracaine was applied topically. The study drug remained on the treatment area for 20-30 minutes for minor dermal procedures and 60 minutes for major dermal procedures
  Other Names: Pliaglis

SUMMARY:
The purpose of this study is to evaluate the safety of one treatment of S-Caine™ Peel (skin numbing cream) applied on healthy skin before a painful dermatologic procedure in adults. This study will also evaluate how well the S-Caine™ Peel eases the pain of the procedure.

DETAILED DESCRIPTION:
The practice of dermatology is seeing a rise in the number of surgical and laser procedures as technological advances have expanded the number of conditions amenable to these evolving therapies. Skin biopsies, shave excisions, deep excisions, electro-surgical procedures, intralesional injections, and laser surgery are frequently performed by dermatologists on a daily basis. Some pain accompanies almost all of these procedures, and a local anesthetic is commonly used. Traditionally, intracutaneous injection of lidocaine (with or without epinephrine) has been the anesthetic of choice. However, patients undergoing these procedures are often afraid of needles and syringes and the pain associated with injections. As a result, topical anesthetic agents have been explored and developed as painless alternatives to injected anesthesia.

S-Caine™ Peel (lidocaine 7% and tetracaine 7% cream) consists of a new eutectic formulation of lidocaine and tetracaine. S-Caine Peel is a topical local anesthetic cream that forms a pliable peel on the skin when exposed to air. S-Caine Peel is not occluded during application.

The purpose of this study is to gain additional safety information for S-Caine Peel when used in minor and major dermal procedures in adults.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older.
* Patient elects to undergo a minor or major dermal procedure.
* Patient is able to read and understand a written informed consent and has signed and dated a written informed consent.

Exclusion Criteria:

* Patient has known allergies, contraindications or sensitivities to lidocaine, tetracaine, or other local anesthetics of the amide or ester type or to any components of the test materials.
* Patient has known active atopic dermatitis at the designated treatment site.
* Patient has damaged, denuded or broken skin at the designated treatment site.
* Patient is pregnant or breastfeeding.
* Patient has participated in an investigational study or clinical trial of an unapproved drug within the previous 30 days.
* Patient has enrolled in any previous study involving S-Caine Peel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2005-05; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 20-30 minutes
  To evaluate the safety of a single administration of S-Caine Peel in providing dermal anesthesia over intact skin prior to a minor and major dermal procedure in adults

SECONDARY OUTCOMES:
Adequacy of Anesthesia | 20-30 minutes
  To evaluate the adequacy of anesthesia provided for the minor and major dermal procedure. The adequacy of anesthesia was evaluated by asking patients whether the study drug provided adequate pain relief for the procedure (yes or no), and by asking the investigator whether the study drug provided adequate anesthesia for the procedure (yes or no).

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Barba, MD, Principal Investigator — International Dermatology Research, Inc.
Locations (5):
- United States (5):
  - International Dermatology Research Inc., Miami, Florida
  - Midwest Cutaneous Research, Clinton Township, Michigan
  - Laser and Skin Surgery Center of New York, New York, New York
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Texas Dermatology Research Institute, Dallas, Texas

REFERENCES:
- See also: Pain — http://www.nlm.nih.gov/medlineplus/pain.html